CLINICAL TRIAL: NCT03337061
Title: A Trial of Mindfulness Meditation for Chronic Insomnia
Acronym: MMI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started - halted by funder
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 174084
Record Dates: First submitted 2017-10-27; First posted 2017-11-08 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Mindfulness) (Experimental): This arm will receive mindfulness-based interventions through a mobile application
  Interventions: Other: Mindfulness Meditation
- Control (Sleep Advice) (No Intervention): This is the control arm that will receive usual care

INTERVENTIONS:
Other: Mindfulness Meditation — Mindfulness Meditation delivered through a mobile application
  Arms: Experimental (Mindfulness)

SUMMARY:
To evaluate the efficacy of mediation therapies on measures of sleep and arousal for people with chronic insomnia and with this the viability of smartphone delivered meditation based approaches at a population level.

DETAILED DESCRIPTION:
Sleep complaints are amongst the commonest in medical practice, and insomnia, the commonest of these affecting transiently 1/3 of the population at some point in the year and 1/3 of this population that is 1 in 10 persisting as chronic insomnia. There are significant consequences on the quality of life for individuals and significant economic burden for society.

Insomnia disorder is characterized as persistent difficulty in falling or staying asleep with resulting daytime dysfunction. Once physical and psychiatric causes have been excluded, current treatment guidelines include pharmacological and behavioural approaches. Hypnotic therapy will reduce sleep latency and increase total sleep time, but there are concerns about drug dependency and side effects (residual day time sleepiness and road traffic accidents and impaired balance). Behavioural treatment (CBTi) has been shown to be effective, but availability is scarce and less than 50% of patients achieve full remission, making alternative approaches desirable.

To optimize availability and to improve outcomes, approaches have included group sessions, single treatment sessions and internet sessions, but these are still limited in the NHS by availability of resources or by expense. Mindfulness meditation, focused non-judgmental awareness and attention on the present moment experience, can promote calmness and relaxation. Several health benefits have been shown across stress related conditions, including sleep disturbance, and its universal availability and ease of application make it an attractive alternative to conventional CBTi.

A randomized controlled trial compared Mindfulness-Based Stress Reduction (MBSR), Mindfulness-Based Therapy for Insomnia (MBTI), and Self-monitoring (SM) in the treatment of chronic insomnia . Results indicate that those receiving mindfulness-based interventions (MBSR or MBTI) had significant reductions in total wake time and pre-sleep arousal from baseline-to-post compared to SM. The study concluded that mindfulness meditation appears to be a viable treatment option for adults with chronic insomnia and could provide an alternative to traditional treatments for insomnia.

A recent meta-analysis of 6 randomised controlled trials demonstrated that mindfulness meditation may contribute to improving sleep in subjects with insomnia compared to a control group. Specifically, mindfulness meditation was found to significantly reduce total wake time, sleep onset latency and sleep quality .

The present study builds upon this work, using a small-scale randomized controlled trial to gather preliminary evidence for the treatment efficacy of a brief mindfulness intervention delivered through a mobile application. Headspace (www.headspace.com) mindfulness app will be used to deliver the meditation content. Headspace currently has over 7 million users worldwide and was recently rated in a systematic review as being the highest quality mindfulness app on the market . Participants are adults with insomnia recruited through a sleep centre, recruited for management of their insomnia.

The potential risks of the study are low, as participants will be exposed to a low dose of mindfulness (10 minutes daily). Adverse effects of meditation have been reported in people with a predisposition to psychiatric illness that underwent extensive mindfulness training, such as a 10-day silent retreat. Negative effects have not been reported from 8-week mindfulness interventions. The benefits from this study include improvement in or resolution of insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Meet the diagnostic criteria for an insomnia disorder. Defined as difficulty initiating or maintaining sleep despite adequate opportunity, with at least one symptom of an associated daytime impairment. Additional quantitative insomnia criteria following research recommendations include frequency (defined as sleep onset latency (SOL) or wake after sleep onset (WASO) > 30 minutes at least 3 nights per week and for chronicity, defined as symptoms lasting > 6 months.
* Have access to an iOS or Android smartphone or a desktop computer with Internet access
* Participants will be required to sign an informed consent form

Exclusion Criteria:

1. Uncontrolled medical condition suspected to interfere with sleep or requiring immediate treatment outside of the study
2. Uncontrolled psychiatric conditions requiring immediate treatment outside of the study, including current major depressive episode
3. Comorbid sleep disorders including obstructive sleep apnea
4. Current use of hypnotic or sedating medications for the purpose of insomnia
5. Inadequate proficiency in English to complete the protocol
6. Participation in other trials concurrently
7. Regular meditation practice defined as equal to or more than 2x weekly for the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia Severity (Insomnia Severity Index) | 8 weeks, 3 and 6 month follow-up
  Insomnia Severity Index (ISI): The Insomnia Severity Index has seven questions. The seven answers are added up to get a total score. This will be administered at baseline, after 8-weeks and at a 3 and 6-month follow-up. The index will be sent to by post and. It will take approximately 5 minutes to complete.
Change in Actigraphy determined wake time (TWT) | 2-week screening, 8-week intervention, 3 and 6-month follow-up
  Actigraphy: Sleep onset latency (SOL) and wake after sleep onset (WASO) will be determined using wrist actigraphy. Participants will be provided with an actiwatch during the screening interview conducted at the beginning of the study. The actiwatch will be worn on the non-dominant arm 24 hours a day, except for while bathing, during the 2-week screening period. Additionally, the actiwatch will be worn for one week after the 8-week intervention and for one week prior to the 3 and 6-month follow-up. Participants will send the actiwatch to the investigator by post after each measurement period. The actiwatch will be sent to participants by post before the next measurement point; apart from the first time point where the participant will be given the actiwatch.

SECONDARY OUTCOMES:
Review of mobile-based mindfulness meditation application for insomnia | 6 months
  Review of use of the mobile application and ascertain it's validity for use within this demographic of patients. The review will be performed using usage of the application by participants over the trial period.
Mindfulness (CAMS-R) | Baseline, 8-weeks, 3 and 6-month follow-up
  Mindfulness Inventory (CAMS-R): The CAMS-R will be administered at baseline, after 8-weeks and at a 3 and 6-month follow-up. The inventory will be sent to participants by post. It will take approximately 5 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Hart, MD, Study Chair — Guys and St Thomas NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No